CLINICAL TRIAL: NCT02985762
Title: A Phase 1, Open-Label Study to Evaluate the Safety and Pharmacokinetics of Local Administration of EXPAREL When Administered for Prolonged Postsurgical Analgesia in Subjects Undergoing Open Spinal Fusion or Reconstructive Surgery
Brief Title: PK Study of EXPAREL in Subjects Undergoing Open Spinal Fusion or Reconstructive Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-117
Record Dates: First submitted 2016-12-02; First posted 2016-12-07 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Spinal Fusion; Pain Management
Keywords: bupivacaine; exparel; analgesic; lumbar spine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EXPAREL 266 mg/20 mL (Other): Eligible subjects, whose surgical incision must be at least 8 cm in length, will receive a single dose of EXPAREL (266 mg/20 mL) expanded in volume with 20-60 mL normal saline, depending on the size of the incision
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL

SUMMARY:
The primary objective of this study is to characterize the pharmacokinetic (PK) profile of EXPAREL when administered via local wound infiltration to subjects undergoing open spinal fusion or reconstructive surgery.

The secondary objectives of this study are to assess the safety, tolerability, and efficacy of EXPAREL in this surgical model.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center, open-label study designed to evaluate the safety and pharmacokinetics of EXPAREL when administered via local wound infiltration to subjects undergoing open cervical or thoracic spinal fusion or reconstructive surgery.

Fifteen subjects are planned for enrollment. Eligible subjects, whose surgical incision must be at least 8 cm in length, will receive a single dose of EXPAREL (266 mg/20 mL) expanded in volume with 20-60 mL normal saline, depending on the size of the incision. Incision will be performed using a posterior surgical approach.

Administration Technique:

Study drug should be injected in the prescribed locations based on the areas of highest nerve density. Study drug will be administered using syringes with 22-gauge needles prior to wound closure. The Investigator must document the size of the incision. Each infiltration site should be spaced 1.0-1.5 cm apart and should deliver approximately 1-1.5 mL into both deep and superficial areas (para-spinous fascia, muscle, and subcutaneous layers). As each incision will have three layers of infiltration, the total volume to be infiltrated can range from 40-80 mL (please refer to below specifics on how to determine total volume of expansion). Following infiltration, the tissue should visibly expand with minimal leakage.

Total Volume of Expansion:

The Investigator must document the total volume used for each surgery.

* EXPAREL (20 mL) + normal saline (20-60 mL based on the incision size) = total volume.
* For example: If the infiltration sites are 1.5 cm apart, then a 10 cm incision would be 10 × 2 sides × 3 layers = 60 cm. If there is 1 mL infiltrated every 1.5 cm, the total volume would be 40 mL.

Screening:

Subjects will be screened within 30 days prior to study drug administration. During the screening visit, which must take place at least 1 day prior to surgery, subjects will be assessed for past or present neurologic, cardiac, and general medical conditions that in the opinion of the Investigator would preclude them from study participation. After the informed consent form (ICF) is signed, a medical/surgical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), neurological assessment, alcohol breath test, urine drug screen, and urine pregnancy test for women of childbearing potential will be conducted.

Trained and qualified Investigators will use their usual standard of care surgical technique to perform the surgery. The use of fentanyl or analogues will be permitted (during surgery only). Intraoperative administration of other opioids or any other analgesic, local anesthetics, or anti-inflammatory agents will be prohibited unless needed to treat an adverse event (AE).

Subjects must remain in the hospital for at least 72 hours after surgery in order to undergo postsurgical assessments. In addition, subjects must return for the 84 hour and 96 hour study assessments.

Day 7 Follow-Up Visit:

All subjects will return on Day 7 for a follow-up visit, which will include vital sign measurements, 12-lead ECG, neurological assessment, blood sample collection for PK analysis, and an AE assessment.

Postsurgical Safety Assessments:

This will include a cardiac assessment (i.e., 12-lead ECG), neurological assessment, and vital signs. Adverse events will be recorded from the time the ICF is signed through Day 30. If a cardiac or neurological AE of special interest or SAE occurs during the study, an unscheduled PK blood sample must be collected. In addition, a 12-lead ECG, vital signs, and any appropriate clinical laboratory tests must be conducted. Cardiac AEs of special interest include chest pain (angina, myocardial infarction), abnormal/irregular heart rate (bradycardia, tachycardia, extrasystoles), and shortness of breath requiring intervention. Neurologic AEs of special interest include altered mental status/altered sensorium, rigidity, dysarthria, seizure, tremors, metallic taste, tinnitus, perioral numbness, visual disturbance, and severe or worsening dizziness. Additionally, the following events are of special interest if they persist or occur beyond 72-hours postdose: dizziness, hyperesthesia, muscular twitching, and tingling/paresthesia.

Postsurgical Efficacy Assessments

Will include pain intensity scores using a 10 cm visual analog scale (VAS) and use of supplemental opioid rescue medication.

Pharmacokinetic Assessment:

Blood samples for PK analysis will be obtained predose (on Day 1 prior to study drug administration); 15 minutes, 30 minutes, 1, 2, 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after the beginning of study drug administration; and on Day 7.

Number of Planned Patients for enrollment is 15 adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age.
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3.
3. Scheduled to undergo primary, ≥3 level cervical or thoracic spine fusion or reconstruction under general anesthesia. The surgical incision must be at least 8 cm in length.
4. Female subject must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
5. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.

Exclusion Criteria:

1. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics or opioids.
2. Contraindication to bupivacaine.
3. Received bupivacaine or any other local anesthetic within 7 days of screening.
4. Receiving workers' compensation.
5. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
6. Non-structural or acute spinal conditions (e.g., cauda equina syndrome, infection, tumor, fracture).
7. Planned concurrent surgical procedure.
8. Comorbidity impacting current physical function or Investigator opinion that it may impact postsurgical rehabilitation.
9. Body weight <50 kg (110 pounds) or a body mass index ≥45 kg/m2.
10. History of coronary or vascular stent placed within the past 3 months (may be extended to 1 year if medically indicated per physician discretion).
11. Have been treated for a deep vein thrombosis, pulmonary embolism, myocardial infarction, or ischemic stroke within the past 6 months (may be extended to 1 year if medically indicated per physician discretion).
12. Severely impaired renal or hepatic function (e.g., serum creatinine level > 2 mg/dL [176.8 μmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN], or serum alanine aminotransferase [ALT] level > 3 times ULN).
13. Any neurologic or psychiatric disorder that might impact postsurgical pain or interfere with study assessments.
14. Malignancy in the last 2 years, per physician discretion.
15. History of misuse, abuse, or dependence on opioid analgesics, other prescription drugs, illicit drugs, or alcohol.
16. Failure to pass the alcohol breath test or urine drug screen.
17. Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postsurgical course.
18. Clinically significant medical or psychiatric disease that, in the opinion of the Investigator, would constitute a contraindication to participation in the study, or cause inability to comply with the study requirements.
19. Received any investigational drug within 30 days prior to study drug administration, and/or has planned administration of another investigational product or procedure during the subject's participation in this study.
20. Previous participation in an EXPAREL study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-versus-time curve from the time of administration extrapolated to infinity. The residual area from the time of the last quantifiable concentration (Ctlast) to infinity is to be calculated using the approximation | 7 days
The VAS pain intensity scores at each assessed timepoint | 72 hours
  Pain intensity scores using the VAS at predose (on Day 1 prior to study drug administration); upon arrival at the post-anesthesia care unit (PACU); at 4, 8, 12, 24, 36, 48, 60, and 72 hours after the beginning of study drug administration; immediately prior to each administration of rescue pain medication; and just prior to hospital discharge
Total inpatient postsurgical opioid consumption (in mg) through 72 hours or hospital discharge | 72 hours
Time to first opioid rescue through 72 hours or hospital discharge | 72 hours
The area under the plasma concentration-versus-time curve from the time of administration to the time of the last quantifiable concentration calculated using the log-linear trapezoidal rule | 7 days
  Pharmacokinetic parameters will be estimated from plasma bupivacaine measurements using non-compartmental analysis, based on the sampling schedule at predose (on Day 1 prior to study drug administration); 15 minutes, 30 minutes, 1, 2, 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96 hours after the beginning of study drug administration; and on Day 7
The maximum observed plasma concentration obtained directly from the experimental data without interpolation. Overall, early Cmax (occurring within 2 hours postdose) and late Cmax (occurring after 2 hours postdose) will be presented | 7 days
The time to maximum plasma concentration (Cmax). Overall, early, and late Tmax will be presented | 7 days
The apparent terminal elimination rate constant determined by log-linear regression of the terminal log-linear segment of the plasma concentration-versus-time curve | 7 days
The apparent terminal elimination half-life calculated as 0.693/λz | 7 days
Incidence of TEAEs through Day 30 | 30 days
Summary of neurological assessments (proportion of subjects who are oriented and proportion of subjects who have any of the neurological events | 30 days
Change from baseline in ECG data closest to the median Tmax | 30 days
Investigator assessment of the ECG (normal, abnormal - not clinically significant, abnormal - clinically significant) | 30 days
Change from baseline in vital signs at each assessed timepoint | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Danesi, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No